CLINICAL TRIAL: NCT04897048
Title: Effect of Short-term Ambulatory Oxygen Therapy on Cardiopulmonary Exercise Capacity in Patients With Interstitial Lung Disease (ILD)
Brief Title: Effect of Short-term Oxygen During CPET in ILD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KEK-ZH-NR. 2012-0251_5
Record Dates: First submitted 2021-05-09; First posted 2021-05-21 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen (Experimental): Supplemental oxygen will be applied via a mask during CPET
  Interventions: Procedure: Incremental exercise test (IET); Procedure: Constant work rate exercise test (CWRET)
- Air (Sham Comparator): Sham ambient air will be applied via mask during CPET
  Interventions: Procedure: Incremental exercise test (IET); Procedure: Constant work rate exercise test (CWRET)

INTERVENTIONS:
Procedure: Incremental exercise test (IET) — Incremental cardio pulmonary exercise test until exhaustion
Procedure: Constant work rate exercise test (CWRET) — constant (on 75% Wmax) cardio pulmonary exercise test until exhaustion

SUMMARY:
In a randomized, sham-controlled crossover trial the investigators will test whether supplemental oxygen given during cardiopulmonary exercise testing will improve exercise performance and physiological parameters in patients with interstitial lung disease.

ELIGIBILITY:
Inclusion Criteria:

* interstitial lung disease, diagnosed by high-resolution CT
* FEV1/FVC >70% and FVC <85% predicted
* stable medication for at least 4 weeks
* Desaturation in SpO2 in 6-minute walk test of ≥ 4% to absolute values ≤ 92%
* Signed Informed Consent
* Male and female patients 18 to 80 years of age

Exclusion Criteria:

* Severe daytime hypoxemia (PaO2 ≤7.3 or <55 mmHg at rest)
* Other clinically significant concomitant disease states (e.g., cardiovascular disease, hepatic dysfunction, etc)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia or confusional state of the subject, neurological or orthopaedic problems with walking disability or inability to ride a bicycle
* Women who are pregnant or breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Work Rate (in watts) | 1 day
  Maximal Work Rate (Watt max) measured during incremental exercise tests (IET) in cardiopulmonary exercise tests
Endurance time (in seconds) | 1 day
  Endurance (sec) with 75% Wmax measured during constant work rate exercise tests (CWRET) in cardiopulmonary exercise tests

SECONDARY OUTCOMES:
changes in physiological vital signs: Heart rate (hr) | 1 day
  Hr (in beats per minute)
changes in physiological vital signs: Blood pressure | 1 day
  Systolic and diastolic blood pressure (in mmHg)
Changes in breathing patterns: Minute ventilation (VE) | 1 day
  VE (in liters per minute)
Changes breathing patterns: Tidal volume (Vt) | 1 day
  Vt (in liters)
Changes in breathing patterns: Oxygen uptake (VO2) | 1 day
  VO2 (in liters per minute)
Changes in breathing patterns: Carbon dioxide output (VCO2) | 1 day
  VCO2 (in liters per minute)
Changes in breathing patterns: Breathing equivalent for O2 (VE/VO2) | 1 day
  ratio between minute ventilation and oxygen uptake
Changes in breathing patterns: Breathing equivalent for O2 (VE/VCO2) | 1 day
  ratio between minute ventilation and carbon dioxide output
Changes in breathing patterns: VE/VCO2Slope | 1 day
  Ratio between minute ventilation and carbon dioxide output if carbon dioxide reaches the breathing plateau
Changes in breathing patterns: Ventilatory threshold one (Vt1) | 1 day
  represents the start of anaerobic metabolism
Changes in breathing patterns: Ventilatory threshold two (Vt2) | 1 day
  represents the start of higher percentage of the anaerobic metabolism
Changes in arterial blood: arterial partial pressure of O2 (PaO2) | 1 day
  PaO2 (in kPa)
Changes in arterial blood: arterial partial pressure of CO2 (PaCO2) | 1 day
  PaCO2 (in kPa)
Changes in arterial blood: arterial lactate concentration | 1 day
  lactate concentration (in mmol per liter)
Changes in arterial blood: pondus Hydrogenii (pH) values | 1 day
  pH (1-14)
Changes in arterial blood: Bicarbonate (HCO3) | 1 day
  HCO3 (in mmol per liter)
Changes in tissue oxygenation: Pulse oxymetrie (SpO2, measured at the finger) | 1 day
  SpO2 (in percent)
Changes in tissue oxygenation: Cerebral tissue oxygenation (CTO, measured at the forehead) | 1 day
  CTO (in percent)
Changes in tissue oxygenation: Muscle tissue oxygenation (MTO, measured at the quadriceps muscle) | 1 day
  MTO (in percent)

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No